CLINICAL TRIAL: NCT00927693
Title: Early Identification of Subclinical Atherosclerosis Using Non-Invasive Imaging Research (EISNER)
Acronym: EISNER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: The Eisner Foundation (Unknown)
Responsible Party: Principal Investigator, Daniel S. Berman, Chief Cardiac Imaging and Nuclear Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3351
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: Atherosclerosis; Coronary Artery Disease; Cardiac Risk Factors; Coronary Calcium Scan; Prevention
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — Carnitine Acyltransferases

ARMS (2):
- Scan group (Experimental): "Scan" group undergoes complete cardiac risk assessment and CAC scanning at baseline.
  Interventions: Other: Coronary Artery Calcium (CAC) Scan
- No scan group (No Intervention): "No scan" group undergoes only complete cardiac risk assessment (without CAC scan) at baseline.

INTERVENTIONS:
Other: Coronary Artery Calcium (CAC) Scan — A coronary artery calcium (CAC) scan is performed during the baseline clinic visit. The results including the actual images from the scan are viewed by the subject during the risk factor consultation with the nurse practitioner. Results are available for the subjects' physicians upon request.
  Arms: Scan group

SUMMARY:
Early Identification of Subclinical Atherosclerosis by Noninvasive Imaging Research (EISNER) is a multi-study research program being conducted at Cedars-Sinai Medical Center.

The principal objective of this randomized trial (referred to as "Study 1") is to assess whether coronary artery calcium (CAC) scanning provides clinical benefit thus improving patient outcomes in asymptomatic subjects with intermediate coronary artery disease (CAD) risk. Additionally, the study is designed to assess the value of combining the CAC scan with the Framingham risk score (FRS) and measurements of serum or plasma biomarkers to predict outcomes.

DETAILED DESCRIPTION:
At baseline eligible subjects underwent a clinic visit where they were randomized 2:1 to a "scan group" which had complete cardiac risk assessment and CAC scanning or a "no scan group" which had only complete cardiac risk assessment. Both groups underwent a private counseling session with a trained nurse practitioner to review their results and receive customized health behavior suggestions based on current American Heart Association guidelines for primary prevention of heart disease.

Subjects were followed up for changes in clinical status, medication use and specific health behaviors at one year after baseline. Annually for four years, subjects were followed up for subsequent diagnostic testing, therapy, and outcomes related to their cardiac health.

At four years after baseline, all subjects (from both groups) returned for a repeat clinic visit to have a complete cardiac risk assessment and CAC scanning. Year 4 CAC scanning was performed in both the "scan group" and "no scan group".

Additional long-term followup is being conducted under a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

* No symptoms of CAD
* Intermediate risk of CAD, defined as either:

  1. male with age of 55-80 years or female with age 65-80 years or
  2. male of 45-54 years and at least one CAD risk factor or female with age 55-64 years and at least one CAD risk factor

     * Risk factors include: smoking, high blood pressure, high total or LDL cholesterol, low HDL cholesterol, diabetes, family history of early CAD.)

Exclusion Criteria:

* History of CVD including heart attack, cardiomyopathy, peripheral artery disease, angina, revascularization, and CVA (stroke)
* Prior coronary calcium scan or coronary angiogram
* Pregnancy
* Required radiation badges for work (CSMC Radiation Safety ruling)
* Clinically unstable health status or significant medical co-morbidity

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2137 (Actual)
Dates: Start 2001-02; Primary Completion 2009-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures include - Coronary artery calcium (CAC) score at Year 4 - CAD risk factors, Framingham Risk Score (FRS), and health behaviors at Year 4 - Adverse cardiac outcomes during follow-up | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Berman, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Lin A, Wong ND, Razipour A, McElhinney PA, Commandeur F, Cadet SJ, Gransar H, Chen X, Cantu S, Miller RJH, Nerlekar N, Wong DTL, Slomka PJ, Rozanski A, Tamarappoo BK, Berman DS, Dey D. Metabolic syndrome, fatty liver, and artificial intelligence-based epicardial adipose tissue measures predict long-term risk of cardiac events: a prospective study. Cardiovasc Diabetol. 2021 Jan 29;20(1):27. doi: 10.1186/s12933-021-01220-x. PMID 33514365
- [Derived] Rozanski A, Gransar H, Shaw LJ, Kim J, Miranda-Peats L, Wong ND, Rana JS, Orakzai R, Hayes SW, Friedman JD, Thomson LE, Polk D, Min J, Budoff MJ, Berman DS. Impact of coronary artery calcium scanning on coronary risk factors and downstream testing the EISNER (Early Identification of Subclinical Atherosclerosis by Noninvasive Imaging Research) prospective randomized trial. J Am Coll Cardiol. 2011 Apr 12;57(15):1622-32. doi: 10.1016/j.jacc.2011.01.019. PMID 21439754